CLINICAL TRIAL: NCT02594787
Title: The Effect of Phosphorus on Diet Induced Thermogenesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lebanese American University (Other)
Responsible Party: Principal Investigator, Maya Bassil, Assistant Professor, Lebanese American University
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: LAU.SOAS.MB1.2012.R1.11
Record Dates: First submitted 2015-11-01; First posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Imbalance of Constituents of Food Intake; Healthy
MeSH Terms: interventions — Phosphorus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phosphorus (Active Comparator): Intervention (500 mg of potassium phosphate) will be administered with 75 g glucose solution and diet induced thermogenesis will be measured afterwards
  Interventions: Dietary Supplement: Phosphorus
- Placebo (Placebo Comparator): Placebo (cellulose) will be administered with 75 g glucose solution and diet induced thermogenesis will be measured afterwards
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Phosphorus
  Arms: Phosphorus
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The aim of the trial is to investigate the effect of ingestion of 75g of glucose (with or without phosphorus) on diet induced thermogenesis (using indirect calorimetry) and appetite (using visual analogue scales) in lean and obese healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Sedentary lifestyle
* Stable weight for the past 3 months
* On a balanced diet

Exclusion Criteria:

* Underweight (BMI<18.5) or overweight/obese (BMI≥25)
* age <18 or > 30 years
* Inability to give valid consent
* Presence of a chronic or acute illness.
* Elevated physical activity level (assesses by the physical activity questionnaire)
* Heavy smokers (≥1 pack per day).
* Weight gain or loss of > 3% in the past 3 months
* History of kidney stones

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2011-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Diet Induced Thermogenesis | 180 minutes (measured every 30 min)
  Diet Induced Thermogenesis will be measured using indirect calorimetry (VO2 consumption)

CONTACTS AND LOCATIONS:
Overall Officials: Maya Bassil, PhD, Principal Investigator — Lebanese American University